CLINICAL TRIAL: NCT04739189
Title: Appetite Response to Exercise- Versus Energy Restriction-induced Energy Deficit in Adolescents With Obesity.
Acronym: IDEX1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Tza Nou - Maison médicale pour enfants et adolescentes (Unknown); Laboratoire AME2P (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2020 JULIAN; 2020-A03567-32 (Other: 2020-A03567-32)
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Pediatric Obesity
Keywords: appetite control; obesity; Adolescents; exercise; Energy Deficit
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese adolescent (Experimental)
  Interventions: Behavioral: Con : control condition without exercise / rest condition; Behavioral: Def-EX : Condition with an exercise-induced energy deficit; Behavioral: Def-EI : Condition with an energy-restriction energy deficit

INTERVENTIONS:
Behavioral: Con : control condition without exercise / rest condition — Control condition without exercise / rest condition. The adolescents will be asked to remain quiet and at rest during the morning and will receive an ad libitum meal at dinner time. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.
Behavioral: Def-EX : Condition with an exercise-induced energy deficit — Condition with an exercise-induced energy deficit The adolescents will be asked to complete an acute exercise set at 65% of their capacities (cycling) during the afternoon, inducing an energy expenditure of 400 kcal. Dinner will be served ad libitum. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.
Behavioral: Def-EI : Condition with an energy-restriction energy deficit — Condition with an energy-restriction energy deficit The adolescents will be asked to remain quiet during the whole day (no physical activity). They will receive a calibrated breakfast reduced from 400 kcal compare to their CON and Def-EX conditions. Dinner will be served ad libitum. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.

SUMMARY:
The aim of the present study is to compare the effect of iso-energetic energy deficits induced by exercise or dietary restriction on energy intake and appetite feelings in adolescents with obesity

DETAILED DESCRIPTION:
The present study will compare the nutritional response to an energy deficit of 400 kcal induced once by realisation of an acute exercise set at moderate intensity and once by a dietary restriction imposed at lunch (compared with a control condition). 18 adolescents with obesity will be asked to randomly complete three experimental sessions: i) one control session (CON); ii) one session with an exercise-induced energy deficit (Def-EX); iii) one session with an energy restriction-induced energy deficit (Def-EI).

Their ad libitum energy intake will be assessed during dinner time. Appetite feelings will be assessed at regular intervals and their food reward in response to the lunch will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI percentile > 97th percentile according to the french curves.
* ages 12-16 years old
* Signed consent form
* being registered in the national social security system
* no contraindication to physical activity

Exclusion Criteria:

* Previous surgical interventions that is considered as non-compatible with the study.
* Diabetes
* weight loss during the last 6 months
* cardiovascular disease or risks

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Change from different intervention of energy intake measured during an ad libitum buffet meal (in kcal) | day 1, day 8, day 15
  food intake will be measured ad libitum during a dinner buffet. The adolescents will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be weighted using an electronic food scale by a member of the investigation team and then analysed using Bilnuts software.

SECONDARY OUTCOMES:
Hunger feelings | day 1, day 8, day 15
  hunger area under the curve will be assessed using visual analogue scale through a the day
Food reward | day 1, day 8, day 15
  The participants will be asked to complete a validated computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie JULIAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moore H, Pereira B, Fillon A, Miguet M, Masurier J, Beaulieu K, Finlayson G, Thivel D. The association between obesity severity and food reward in adolescents with obesity: a one-stage individual participant data meta-analysis. Eur J Nutr. 2024 Jun;63(4):1241-1255. doi: 10.1007/s00394-024-03348-4. Epub 2024 Feb 20. PMID 38376518